CLINICAL TRIAL: NCT01397032
Title: Attention Bias Modification Treatment for Children With Social Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Head of Shcool of Psychological Sciences, Tel-Aviv University, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2009340
Record Dates: First submitted 2011-06-20; First posted 2011-07-19 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Social Phobia
Keywords: attention bias modification treatment; cognitive bias modification; attention training; social anxiety
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification (ABM) (Experimental): Attention training via repeated trials of a dot-probe task intended to direct attention away from threat stimuli.
  Interventions: Behavioral: Attention Bias Modification Treatment (ABMT)
- Placebo (Placebo Comparator): Attention training via repeated trials of a dot-probe task not intended to change threat-related attention patterns.
  Interventions: Behavioral: Attention Control Condition

INTERVENTIONS:
Behavioral: Attention Bias Modification Treatment (ABMT) — Behavioral: Attention Bias Modification Treatment (ABMT) Attention training using a computerized spatial attention task (dot-probe) modified to alter threat-related attention patterns.
  Arms: Attention Bias Modification (ABM)
Behavioral: Attention Control Condition — Attention training using a computerized spatial attention task (dot-probe) not intended to alter threat-related attention patterns.
  Arms: Placebo

SUMMARY:
Children with social anxiety will be randomly assigned to either Attention Bias Modification Treatment (ABMT) designed to direct attention away from threat or a placebo control condition not designed to change attention patterns. Outcome measures will be depression and social anxiety symptoms as measured by gold standard questionnaires as well as diagnosis of social phobia disorder and symptom counts derived from structured clinical interviews with children and their parents.

We expect to see significant reduction in social anxiety symptoms in the Attention Bias Modification Treatment (ABMT) group relative to the placebo control group.

ELIGIBILITY:
Inclusion Criteria:

* children suffering from social anxiety

Exclusion Criteria:

* Pharmacological or Psychological treatment

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2011-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV (ADIS) | expected average time frame of 6 weeks. Participants will be assessed before and after the administriation of the training/control protocols.
  The ADIS is a semi-structured interview assessing anxiety, mood and externalizing disorders in children according to DSM-IV criteria.

SECONDARY OUTCOMES:
Social Phobia and Anxiety Inventory for Children (SPAI-C) and for Parents (SPAI-c-p) | expected average time frame of 6 weeks. Participants will be assessed before and after the administriation of the training/control protocols.
  The SPAI is a 26-item self and parent-report instrument designed to assess social anxiety in children and adolescents. Items assess a range of potentially anxiety-producing situations.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel

REFERENCES:
- [Background] Hakamata Y, Lissek S, Bar-Haim Y, Britton JC, Fox NA, Leibenluft E, Ernst M, Pine DS. Attention bias modification treatment: a meta-analysis toward the establishment of novel treatment for anxiety. Biol Psychiatry. 2010 Dec 1;68(11):982-90. doi: 10.1016/j.biopsych.2010.07.021. PMID 20887977
- [Derived] Pergamin-Hight L, Pine DS, Fox NA, Bar-Haim Y. Attention bias modification for youth with social anxiety disorder. J Child Psychol Psychiatry. 2016 Nov;57(11):1317-1325. doi: 10.1111/jcpp.12599. Epub 2016 Jul 20. PMID 27435286